## SimuVersity Medical Center: Pain and Opioid Management Training in Diverse Patient Populations

Informed Consent Form

NCT06624124

March 10, 2025

## Volunteer Statement

If you are a faculty member or student at the Medical University of South Carolina between the ages of 18 and 80, you are eligible to volunteer to participate in a research study looking at the impact of a new game-based technology to teach health professionals about pain management and diversity considerations in health care. The Principal Investigator of this study is Dr. Jeff Borckardt.

Your participation is online and self-paced and will take 1 to 2 hours. During participation, you will interact with online training materials and review clinical case studies. You will be randomly assigned (50/50 chance; like a coin flip) to either learn about pain management and diversity through a video-game-like interface and practice applying knowledge using digital/virtual patients -OR- by viewing powerpoint slides and reviewing text-based case studies.

You will be asked about your degree program, age, sex, race and ethnicity, video game experience, and complete pre- and post-training knowledge tests as well as rating scales about your experience with the learning activity.

While loss of confidentiality is always a risk in research studies, the research team has put safeguards in place to ensure that your personal information is protected and that there is no loss of confidentiality.

Upon completion of the training activity you will be prompted to enter your email address and the Office of Interprofessional Initiatives front desk will email you a link to a \$30 Amazon gift card. Your email address will not be linked with your study data. It will be provided for renumeration purposes only.

Your participation is voluntary and your participation or discontinuance will not impact any element of your job or educational performance/evaluation and will not become a part of your student or employment record.

Choosing to participate in the project implies your understanding and willingness to participate.

If you have any questions, Please contact Dr. Borckardt at borckard@musc.edu



IRB Number: Pro00137370 Date Approved 3/10/2025

Changing What's Possible